CLINICAL TRIAL: NCT01243788
Title: Efficacy and Safety of Salmeterol/Fluticasone Propionate vs Ipratropium/Albuterolin Chinese Patients With Moderate-to-severe COPD.
Brief Title: The Efficacy and Safety of Salmeterol/Fluticasone Propionate vs Atropium/Albuterol in Patients COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Guangzhou First People's Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Chao Yang Hospital (Other); Peking University Third Hospital (Other); Liaoning Cancer Hospital & Institute (Other); West China Hospital (Other); Xinqiao Hospital of Chongqing (Other); Qingdao University (Other); Armed Police Medical college Affiliated Hospital (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Chunxue BAI, Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCO113162; SCO113162 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Seretide; Combivent; effect and safety; Twelve weeks
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipratropium/Albuterol (Active Comparator): Ipratropium/Albuterol 36/206ug QID
  Interventions: Drug: Salmeterol/Fluticasone Propionate

INTERVENTIONS:
Drug: Salmeterol/Fluticasone Propionate — Salmeterol/Fluticasone 50/500ug twice daily Duration:12 weeks
  Other Names: Combivent; Salbutamol Aerosol

SUMMARY:
To determine the efficacy and safety of Salmeterol/Fluticasone Propionate 50/500ug BID vs Ipratropium/Albuterol 36/206ug QID in Chinese patients with moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
* This is a 12-week, multicentre,randomized,open-label,active-controlled, paralleled-group study.
* Chinese patients aged ≥40 years with moderate-to-severe COPD are eligible for this study.

  1. If satisfying the entry criteria, patients enter an 8 to 14 day run-in period,and replace previous bronchodilators with inhaled or nebulized Salbutamol.
  2. Patients record daily severity ratings for daytime symptoms of shortness of breath, tiredness, activity limitation, frustration with symptoms, and night-time sleep symptoms on daily cards.
  3. Each symptom is rated using 0-100 visual analog scal (VAS). For overall assessment of daytime symptoms, a combined symptom score is obtained by adding VAS scores for shortness of breath, tiredness, activity limitation, frustration with symptoms.
  4. Patients are required to be symptomatic as demonstrated by a combined daytime symptom score of 120 on at least 4 of the 7 days prior to randomization.

  <!-- -->

  1. Eligible patients will be randomized (1:1) to the following 2 treatments for 12 weeks.

     1. Inhaled Salmeterol/Fluticasone propionate 50/500ug twice daily or inhaled IB/ALB 36/206ug QID.
     2. Salbutamol will be provided for relief of symptoms on an "as required" basis during the whole 12 weeks.
  2. A Follow-up visit will be conducted 2 weeks after completion of treatment/early withdrawal to assess for any adverse effects after discontinuing study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female outpatients aged 40 to 79 years, inclusive
* Patients with an established diagnosis of COPD, defined as GOLD guideline postbronchodilation FEV1/FVC ratio of <70%, AND Postbronchodilation FEV1% predicted ranged from ≥25 to ≤70.
* A cigarette smoking history of 10 pack-years
* Use of oral theophylline, or any other inhaled medications other than LABA, LAMA, or ICS for≥30 days (e.g. SABA, SAMA)
* Patients who are able to use Accuhaler device and relief medication
* Patients willing to give informed consent to participate in the study and comply to study protocol
* Eligible female on child-bearing potentia

Exclusion Criteria:

* Patients with concurrent respiratory disorders (e.g. asthma) other than COPD
* Patients with a requirement for regular or long term oxygen therapy (>12h/d)
* Patients who used inhaled or oral steroids within 30 days of screening
* Patients who had a respiratory tract infection requiring antibiotics within 14 days of screening
* Patients with a moderate-to-severe COPD exacerbation within 30 days of screening
* Patients with any significant medical condition or disease that would place patients at risk or interfere with the study evaluation.
* Patients who used some inhibitory agents (e.g. b blockers) within 14 days of screening
* Female patients who is pregnant or may be pregnant in the study duration

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-02 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
pre-broncholidator FEV1 | at 12 weeks
  Change from Baseline in pre-broncholidator FEV1 at 12 weeks

SECONDARY OUTCOMES:
post-broncholidator FEV1 | at 12 weeks
  Change from Baseline in post-broncholidator FEV1 at 12 weeks
Morning PEF, inspiration capacity (IC) and Residual Volume (RV) | at 12 weeks
  Change from Baseline in morning PEF, inspiration capacity (IC) and Residual Volume (RV)at 12 weeks
Overall daytime symptom score, reliever medication use,SGRQ and BODY index | at 12 weeks
  Change from Baseline in overall daytime symptom score, reliever medication use,SGRQ and BODY index at 12 weeks
Percent of symptom-free nights, sleep symptoms, nighttime awakenings due to respiratory symptoms | at 12 weeks
  Change from Baseline in percent of symptom-free nights, sleep symptoms, nighttime awakenings due to respiratory symptoms at 12 weeks
Biomarkers: serum Clara cell 16 (CC-16) protein and serum surfactant protein D (SPD) | at 12 weeks
  Change from Baseline in biomarkers: serum Clara cell 16 (CC-16) protein and serum surfactant protein D (SPD) at 12 weeks
participants with adverse events and COPD exacerbations | at 12 weeks
  Change from Baseline in number of participants with adverse events and COPD exacerbations at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue C BAI, Doctor, Principal Investigator — Fudan University
Locations (11):
- China (11):
  - Affiliated Hospital of Anhui Medical College, Hefei, Anhui
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Gguang Zhou Institute of Respiratory Disease, Guangzhou, Guangdong
  - Henan Province Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital,, Wuxi, Jiangsu
  - Shenyang Military General Hospital, Shenyang, Liaoning
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan, Chengdu, Sichuan
  - Chongqing Xinqiao Hospital, Chongqing, Sichuan